CLINICAL TRIAL: NCT03141086
Title: A Randomized, Subject and Investigator-blinded, Placebo Controlled, Cross-over, Multi-center Proof of Concept (PoC) Study to Assess the Wakefulness Promoting Effect, Safety, Tolerability, and PK of LML134 in Shift Work Disorder (SWD) Patients
Brief Title: A Study to Assess the Wakefulness Promoting Effect, Safety, Tolerability, and Pharmacokinetics (PK) of LML134 in Shift Work Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CLML134X2201 was terminated due to business reasons and not to safety findings
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLML134X2201
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Results first posted 2019-09-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-06

CONDITIONS: Circadian Rhythm Disorders
Keywords: shift work disorder
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): LML134, then placebo
  Interventions: Drug: LML134; Drug: Placebo
- Group 2 (Experimental): Placebo, then LML134
  Interventions: Drug: LML134; Drug: Placebo

INTERVENTIONS:
Drug: LML134 — LML134
Drug: Placebo — placebo

SUMMARY:
The main purpose of this study was to demonstrate that LML134 can increase wakefulness compared to placebo in patients with shift work disorder (SWD) measured by objective and subjective endpoints of wakefulness, i.e. the sleep latency in the multiple sleep latency test (MSLT) and the Karolinska Sleepiness Scale (KSS), respectively. Safety and PK of LML134 were also evaluated. In addition, novel methodologies to measure wakefulness and sleep were also to be tested and compared to gold standard methods like the MSLT and polysomnography (PSG) (at sites where staff have appropriate equipment and training). The aim of such comparisons was to evaluate the usefulness of the new technologies in clinical studies and provide preliminary validation data.

This was a randomized, subject and investigator-blinded, placebo controlled, crossover, multi-center Proof of Concept (PoC) study with in-house simulated laboratory night shifts in patients with SWD. This non-confirmatory study included two treatment arms: LML134 and placebo. After a screening period, the treatment phase of the study consisted of two overnight stays in a sleep lab in each of two treatment periods, with a minimum one week wash-out in between.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 65 years of age included.
* Confirmed diagnosis of SWD according to ICSD-3 criteria at Screening.
* Subjects who are at least moderately ill with respect to sleepiness on work nights, including commute to and from work, as assessed by the Clinical Global Impression-Severity scale (CGI-S, score ≥4) at Screening.
* Subjects must work 5 or more night shifts per month, and 2 or more shifts must occur on consecutive nights, with 6 or more hours worked between 10 pm and 8 am, as confirmed by subject at Screening.
* Subjects must have mean sleep latency ≤8 minutes on nighttime MSLT at Screening.
* Subjects must weigh at least 50 kg at Screening to participate in the study, and must have a body mass index (BMI) within the range of 18 - 35 kg/m2. BMI = Body weight (kg) / [Height (m)]2

Exclusion Criteria:

* Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) unless they are using highly effective methods of contraception from start of taking the study medication in the first period until stopping the medication in the second treatment period and for 3 additional days after AND an additional barrier method of contraception will be used while taking the study medication and for 3 additional days in both treatment periods.
* Sexually active males unwilling to use a condom during intercourse while taking investigational drug and for 3 days after stopping investigational drug. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of the investigational drug via seminal fluid to their partner.
* Heavy smokers who smoke more than 10 cigarettes a day and occasional or light smokers (not more than 10 cigarettes per day) who are not willing to, or in their own or the investigators opinion are not able to refrain from tobacco/nicotine use for at least 12 hours without nicotine craving or other withdrawal symptoms
* Subjects for whom it is not safe to discontinue or who are unwilling to discontinue use of modafinil, hypnotics, and antihistamines for the periods specified in the prohibited medication section.
* Heavy caffeine consumers, i.e. subjects who consume greater than 850 mg of caffeine per day (approximate equivalent of three tall cups of Starbucks coffee) in coffee, tea, or other caffeine-containing drinks.
* Subjects who have high risk of obstructive sleep apnea, indicated by score of 5 or more on the STOP-BANG questionnaire.
* Presence of any sleep disorder other than SWD, as confirmed by PSG at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Oakland Park, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chevy Chase, Maryland
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Originally 46 subjects were planned to be enrolled in the study. However, 24 subjects were actually enrolled in the study and randomized as the study was prematurely terminated for business reasons.
Groups:
- Group 1: LML134, Then Placebo: LML134, then placebo
- Group 2: Placebo, Then LML134: Placebo, then LML134
Period: Overall Study
Arm/Group | Group 1: LML134, Then Placebo | Group 2: Placebo, Then LML134
Started | 7 | 17
Completed | 6 | 12
Not Completed | 1 | 5
Not completed — Study Terminated By Sponsor | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: LML134, Then Placebo | Group 2: Placebo, Then LML134 | Total
Number analyzed (Participants) | 7 | 17 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.0 (10.42) | 39.3 (10.00) | 40.7 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 6 | 14 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 6 | 6 | 12
  White | 1 | 11 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Sleep Latency Over Two Consecutive Test Nights as Measured by the the Multiple Sleep Latency Test (MSLT)
Description: The Multiple Sleep Latency Test (MSLT) is an objective assessment of sleepiness that measures the ability of a subject to remain awake. Long latencies to sleep are indicative of a patient's ability to remain awake. Mean sleep latency from MSLT was measured for four MSLT naps performed at scheduled timepoints (01:30, 03:30, 05:30, and 07:30). The primary efficacy variable was the mean MSLT sleep latency assessed at Day 1 and Day 2 of each treatment period.
Time Frame: Day 1 and Day 2 of each treatment period (midnight until 8:00)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: min
Groups:
- LML134 5mg: LML134 5mg
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 20 | 23
min | 6.76 (4.154) | 4.12 (2.993)
Statistical Analysis 1: Comparison: LML134 5mg vs Placebo; Test type: Superiority; p = 0.1272, ANOVA; Mean Difference (Final Values) = 1.711, 95% CI 2-sided [-1.340 to 4.762]

2. Secondary Outcome: Sleep Latency at Separate Naps Over Two Consecutive Test Nights as Measured by the the Multiple Sleep Latency Test (MSLT)
Description: The Multiple Sleep Latency Test (MSLT) is an objective assessment of sleepiness that measures the ability of a subject to remain awake. Long latencies to sleep are indicative of a patient's ability to remain awake. Mean sleep latency from MSLT was measured for four MSLT naps performed at scheduled timepoints (01:30, 03:30, 05:30, and 07:30). The outcome measure is the mean value of Day 1 and Day 2 assessments for each timepoint.
Time Frame: Day 1 and Day 2 of each treatment period (midnight until 8:00)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 20 | 23
min
  01:30 (3.5 hours post dose) | 8.73 (6.191) | 5.27 (5.065)
  03:30 (5.5 hours post dose) | 7.13 (5.188) | 4.57 (4.494)
  05:30 (7.5 hours post dose) | 5.18 (5.160) | 3.38 (3.398)
  07:30 (9.5 hours post dose): number analyzed (Participants) | 19 | 23
  07:30 (9.5 hours post dose) | 5.29 (4.772) | 3.25 (2.726)
Statistical Analysis 1: Comparison: LML134 5mg vs Placebo; 3.5 hours post dose; Test type: Superiority; p = 0.0607, Mixed Models Analysis; Mean Difference (Final Values) = 2.866, 95% CI 2-sided [-0.821 to 6.553]
Statistical Analysis 2: Comparison: LML134 5mg vs Placebo; 5.5 hours post dose; Test type: Superiority; p = 0.0919, Mixed Models Analysis; Mean Difference (Net) = 1.975, 95% CI 2-sided [-1.024 to 4.973]
Statistical Analysis 3: Comparison: LML134 5mg vs Placebo; 7.5 hours post dose; Test type: Superiority; p = 0.0811, Mixed Models Analysis; Mean Difference (Net) = 1.576, 95% CI 2-sided [-0.697 to 3.848]
Statistical Analysis 4: Comparison: LML134 5mg vs Placebo; 9.5 hours post dose; Test type: Superiority; p = 0.2026, Mixed Models Analysis; Mean Difference (Net) = 0.879, 95% CI 2-sided [-1.268 to 3.026]

3. Secondary Outcome: Plasma PK Concentration
Description: Plasma PK concentration. Due to sparse sampling, only plasma concentrations were calculated and no PK parameter was evaluated by non-compartmental analysis.
Time Frame: 0 to 34.5 hours post first treatment.
Population: Pharmacokinetic analysis set (only analyzed for LML134 treatment period - not analyzed for Placebo period)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LML134 5mg
Number analyzed (Participants) | 21
ng/mL
  pre-dose | 0 (0)
  0.25 hours post dose | 0.184 (0.406)
  3 hours post dose | 24.1 (11.3)
  12 hours post dose: number analyzed (Participants) | 20
  12 hours post dose | 6.53 (5.25)
  24 hours post dose: number analyzed (Participants) | 19
  24 hours post dose | 1.31 (1.59)
  34.5 hrs post 1st dose (10.5 hrs post 2nd dose): number analyzed (Participants) | 19
  34.5 hrs post 1st dose (10.5 hrs post 2nd dose) | 7.55 (5.72)

4. Secondary Outcome: Total Time in Bed Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Total time in bed is the time spent in bed during recording.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
min | 479.9 (0.16) | 480.0 (0.14)

5. Secondary Outcome: Sleep Time Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Total sleep time is the overall duration of sleep during the entire PSG recording.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
min | 253.8 (102.53) | 294.8 (87.94)

6. Secondary Outcome: Sleep Efficiency Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Sleep efficiency is the percentage of time spent asleep during the entire PSG recording.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
percentage of time | 53.1 (21.17) | 61.4 (18.32)

7. Secondary Outcome: Wake Time After Persistent Sleep Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Wake time after persistent sleep is a measure of time spent awake after a defined onset of sleep.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
min | 214.9 (101.88) | 174.2 (87.48)

8. Secondary Outcome: Latency to Onset of Persistent Sleep Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep. Latency to onset of persistent sleep is defined as latency from Lights-Off to the first epoch (30 seconds) of 20 consecutive epochs of non-Wake.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
min | 8.1 (8.92) | 11.0 (12.63)

9. Secondary Outcome: Number of Awakenings Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Number of awakenings is defined as the number of times of entering wake stage after onset of sleep during the PSG recording.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
awakenings | 11.7 (5.29) | 12.2 (7.45)

10. Secondary Outcome: Latency to Rapid Eye Movement (REM) Sleep Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Sleep latency to REM Sleep is defined as the time from Lights-Off to reaching the first epoch (i.e. 30 seconds) of REM sleep.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
min | 89.7 (53.09) | 44.9 (38.05)

11. Secondary Outcome: Number of Sleep Cycles Measured by Polysomnography (PSG)
Description: PSG encompasses the monitoring of subjects in a sleep facility using an array of medical equipment with simultaneously recording on a multi-channel analog or digital system. PSG was performed in the study to record and evaluate various aspects of sleep.
  Number of sleep cycles measured by Polysomnography (PSG).
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis set - this outcome measure was not recorded in the Polysomnography testing
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Time Spent in Each Sleep Stage Measured by Polysomnography (PSG)
Description: N1: is defined by a relatively low amplitude, mixed frequency EEG. N2: is defined by the presence of sleep spindles and/or K complexes and the absence of sufficient high-amplitude, slow activity to define the presence of stage N3 sleep.
  N3: is defined as an EEG with at least 20% of an epoch consisting of slow, high amplitude waveforms of .5 - 2 Hz and peak-to-peak amplitude of greater than 75mV.
  REM: is defined by the concomitant appearance of relatively low amplitude, mixed frequency EEG activity and episodes of rapid eye movement. Sawtooth waves may be present. Chin EMG activity is typically low.
Time Frame: Day 2 (10:00 until 18:00) of each treatment period
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: min
Arm/Group | LML134 5mg | Placebo
Number analyzed (Participants) | 19 | 23
min
  N1 | 21.6 (13.95) | 25.1 (16.37)
  N2 | 145.7 (55.68) | 155.2 (58.84)
  N3 | 43.6 (32.70) | 51.1 (29.99)
  REM | 42.9 (30.21) | 63.3 (26.52)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 24 days from first dose of study treatment in each treatment period.
Arm/Group | LML134 5mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 5/21 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LML134 5mg (N=21) | Placebo (N=23)
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03141086/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03141086/SAP_001.pdf